CLINICAL TRIAL: NCT07393217
Title: Circulating Fibroblast Activation Protein (FAP) As A Marker for Fibroblast-Driven Pathology in Rheumatoid Arthritis and Systemic Sclerosis : Implication for Joint, Skin and Lung Fibrosis
Brief Title: Correlation Between Circulating Fibroblast Activation Protein (FAP) and Fibrosis in Two Diseases (Rheumatoid Arthritis and Systemic Sclerosis)
Acronym: FAP
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Toqa Mahfouz Mohamed Ahmed, assistant lecturer at Rheumatology department, Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med--25-12-9MD
Record Dates: First submitted 2026-01-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA); Systemic Sclerosis (SSc)
Keywords: Fibroblast Activation protein; Rheumatoid Arthritis; systemic sclerosis; lung fibrosis; skin fibrosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Scleroderma, Systemic; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Rheumatoid arthritis patients
- systemic sclerosis patients
- control healthy group

SUMMARY:
This study aims to measure a blood protein called fibroblast activation protein (FAP), which is linked to tissue scarring and inflammation. A small blood sample will be taken from participants (RA , SSc patients and healthy people ), and the FAP level will be measured and compared with routine clinical examinations, imaging studies, and lung function tests.

The purpose of this study is to improve understanding of disease activity and lung involvement in these conditions and to explore whether FAP could be useful as a blood marker for future patients. Participation in this study will not change the participant's usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years. Confirmed diagnosis of RA (ACR/EULAR) or SSc (ACR/EULAR).
* Ability and willingness to provide informed consent. Cooperative patient able to answer questions.

Exclusion Criteria:

* Patients under 18 years' old
* Active cancer or history of cancer within 5 years.
* Other major fibrotic systemic disease that could confound circulating FAP levels.
* Acute infection at time of sampling.
* Pregnancy or breastfeeding.
* Other autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients diagnosed with rheumatoid arthritis (RA) or systemic sclerosis (SSc). Participants will be recruited consecutively from the Rheumatology and Rehabilitation outpatient clinics and inpatient units of the study center.
  The sample will consist of three parallel groups:
  Patients with rheumatoid arthritis diagnosed according to the 2010 ACR/EULAR classification criteria.
  Patients with systemic sclerosis diagnosed according to the 2013 ACR/EULAR classification criteria.
  Healthy population who don't have any autoimmune disease.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Serum fibroblast activation protein (FAP) concentration measured by ELISA in patients with rheumatoid arthritis and systemic sclerosis | At baseline (Day 1)

SECONDARY OUTCOMES:
disease activity | baseline
  Correlation between serum FAP concentration and disease activity score in rheumatoid arthritis and systemic sclerosis
pulmonary involvement | baseline
  Correlation between serum FAP concentration and pulmonary involvement in patients with rheumatoid arthritis and systemic sclerosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided